CLINICAL TRIAL: NCT02606487
Title: Hyperpolarized Xenon MRI in Cystic Fibrosis Pulmonary Exacerbations
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Felix Ratjen, Division Head, Respiratory Medicine, The Hospital for Sick Children
Other Study IDs: 1000049033
Record Dates: First submitted 2015-11-13; First posted 2015-11-17 (Estimated); Last update posted 2018-10-04 (Actual); Status verified 2018-10

CONDITIONS: Cystic Fibrosis
Keywords: CF; Exacerbation; Hyerpolarized xenon MRI; Pediatrics; Lung Clearance Index
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CF pulmonary exacerbation group: Patients with cystic fibrosis admitted for inpatient treatment of a pulmonary exacerbation

SUMMARY:
The investigators aim to assess whether pulmonary MRI (hyperpolarised 129Xe ventilation imaging [Xe-MRI]) can detect changes in ventilation defects in patients with CF before and after treatment for a pulmonary exacerbation. The investigators will determine whether changes seen using pulmonary Xe-MRI are associated with changes in pulmonary function (spirometry, lung volumes, lung clearance index [LCI]) in patients with CF before and after pulmonary exacerbation.

DETAILED DESCRIPTION:
Cystic fibrosis (CF) is one of the most common genetic diseases affecting children and young adults [1]. Lung disease is the primary cause of morbidity and mortality in these patients and sensitive markers of lung disease in CF are important for directing therapy in these patients.

LCI, measured by multiple breath washout (MBW), has been shown to be more sensitive than traditional pulmonary function tests (PFTs) for assessing the treatment effect of novel therapies in CF patients [2,3]. However, LCI provides no information regarding the spatial distribution of ventilation inhomogeneity within the lungs and improvements in mucus plugging of poorly ventilated regions can paradoxically worsen the LCI [4,5]. Thus an imaging technique that can capture regional changes in the distribution of ventilation might be better suited than LCI to detect treatment effects and could also help to better define the utility of LCI as a clinical tool.

Xe-MRI is a safe, non-ionizing modality for imaging the lungs, providing an accurate spatial representation of ventilation inhomogeneity [6]. Xe-MRI has been shown to be effective in imaging of adult patients with chronic obstructive pulmonary disease (COPD) and CF [6] however, there are no published studies using Xe-MRI in children.

The hypothesis of this study is that Xe-MRI and LCI will provide complimentary information when quantifying ventilation inhomogeneity in CF lung disease and that Xe-MRI will be able to define patients in whom LCI fails to capture positive effects of treatment. The ultimate goal is to develop more sensitive tools for longitudinal monitoring to direct the clinical care of CF patients in the future.

To accomplish this, the investigators will compare the ability of Xe-MRI and LCI to detect changes in ventilation inhomogeneity in patients with CF before and after treatment for a pulmonary exacerbation, a common pulmonary complication of CF.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CF as defined by two or more clinical features of CF and a documented sweat chloride > 60mEq/L by quantitative pilocarpine iontophoresis test or a genotype showing two well characterized disease causing mutations
* Informed consent and verbal assent (as appropriate) provided by the subject's parent or legal guardian and the subject
* Ages 8-18 years and able to perform reproducible spirometry and achieve a breath hold duration sufficient for MRI acquisition
* Admission to the Hospital for Sick Children for a pulmonary exacerbation (based on clinical or pulmonary function assessment). Children who will be admitted and then discharged on home IV antibiotics may also be included in this study.

Exclusion Criteria:

* Inability to perform reproducible pulmonary function tests (spirometry, plethysmography or lung clearance index) or perform a breath-hold of sufficient duration for MRI acquisition
* Medical instability that would preclude the ability to undergo the required investigations
* FEV1 % predicted < 40%
* Use of supplementary oxygen
* Severe claustrophobia
* Pregnancy or lactation
* Presence of metal implants or other contraindications to MRI

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients aged 8-18 with cystic fibrosis admitted for inpatient treatment with a clinical diagnosis of pulmonary exacerbation
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2015-11; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Ventilation Defect Percentage (VDP) | Pre-treatment
  VDP within 48h of initiation of inpatient treatment
Ventilation Defect Percentage (VDP) | Post-treatment - within 48h of completion of inpatient treatment
  VDP within 48h of completion of inpatient treatment
Lung Clearance Index (LCI) | Pre-treatment
  LCI within 48h of initiation of inpatient treatment
Lung Clearance Index (LCI) | Post-treatment - within 48h of completion of inpatient treatment
  LCI within 48h of completion of inpatient treatment

SECONDARY OUTCOMES:
Pulmonary function tests (PFTs) | Pre-treatment
  PFTs within 48h of initiation of inpatient treatment
Pulmonary function tests (PFTs) | Post-treatment - within 48h of completion of inpatient treatment
  PFTs within 48h of completion of inpatient treatment

CONTACTS AND LOCATIONS:
Overall Officials: Felix Ratjen, MD PhD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Background] O'Sullivan BP, Freedman SD. Cystic fibrosis. Lancet. 2009 May 30;373(9678):1891-904. doi: 10.1016/S0140-6736(09)60327-5. Epub 2009 May 4. PMID 19403164
- [Background] Robinson PD, Latzin P, Verbanck S, Hall GL, Horsley A, Gappa M, Thamrin C, Arets HG, Aurora P, Fuchs SI, King GG, Lum S, Macleod K, Paiva M, Pillow JJ, Ranganathan S, Ratjen F, Singer F, Sonnappa S, Stocks J, Subbarao P, Thompson BR, Gustafsson PM. Consensus statement for inert gas washout measurement using multiple- and single- breath tests. Eur Respir J. 2013 Mar;41(3):507-22. doi: 10.1183/09031936.00069712. Epub 2013 Feb 8. PMID 23397305
- [Background] Davies J, Sheridan H, Bell N, Cunningham S, Davis SD, Elborn JS, Milla CE, Starner TD, Weiner DJ, Lee PS, Ratjen F. Assessment of clinical response to ivacaftor with lung clearance index in cystic fibrosis patients with a G551D-CFTR mutation and preserved spirometry: a randomised controlled trial. Lancet Respir Med. 2013 Oct;1(8):630-638. doi: 10.1016/S2213-2600(13)70182-6. Epub 2013 Sep 10. PMID 24461666
- [Background] Horsley AR, Davies JC, Gray RD, Macleod KA, Donovan J, Aziz ZA, Bell NJ, Rainer M, Mt-Isa S, Voase N, Dewar MH, Saunders C, Gibson JS, Parra-Leiton J, Larsen MD, Jeswiet S, Soussi S, Bakar Y, Meister MG, Tyler P, Doherty A, Hansell DM, Ashby D, Hyde SC, Gill DR, Greening AP, Porteous DJ, Innes JA, Boyd AC, Griesenbach U, Cunningham S, Alton EW. Changes in physiological, functional and structural markers of cystic fibrosis lung disease with treatment of a pulmonary exacerbation. Thorax. 2013 Jun;68(6):532-9. doi: 10.1136/thoraxjnl-2012-202538. Epub 2013 Feb 9. PMID 23396354
- [Background] Yammine S, Bigler A, Casaulta C, Singer F, Latzin P. Reasons for heterogeneous change in LCI in children with cystic fibrosis after antibiotic treatment. Thorax. 2014 Feb;69(2):183. doi: 10.1136/thoraxjnl-2013-204283. Epub 2013 Aug 29. No abstract available. PMID 23988751
- [Background] Shukla Y, Wheatley A, Kirby M, Svenningsen S, Farag A, Santyr GE, Paterson NA, McCormack DG, Parraga G. Hyperpolarized 129Xe magnetic resonance imaging: tolerability in healthy volunteers and subjects with pulmonary disease. Acad Radiol. 2012 Aug;19(8):941-51. doi: 10.1016/j.acra.2012.03.018. Epub 2012 May 15. PMID 22591724
- [Derived] Munidasa S, Couch MJ, Rayment JH, Voskrebenzev A, Seethamraju R, Vogel-Claussen J, Ratjen F, Santyr G. Free-breathing MRI for monitoring ventilation changes following antibiotic treatment of pulmonary exacerbations in paediatric cystic fibrosis. Eur Respir J. 2021 Apr 15;57(4):2003104. doi: 10.1183/13993003.03104-2020. Print 2021 Apr. No abstract available. PMID 33303537